CLINICAL TRIAL: NCT00965328
Title: Nadroparin Anticoagulation for Continuous Venovenous Hemofiltration (CVVH), a Randomized Cross-over Trial Comparing Hemostasis Between Two Hemofiltration Rates
Brief Title: Nadroparin Anticoagulation for Continuous Venovenous Hemofiltration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: HM Oudemans-van Straaten, Onze Lieve Vrouwe Gasthuis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: WO 06044
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Kidney; Acute Renal Failure; Multiple Organ Failure
Keywords: anticoagulation; hemofiltration; acute kidney injury; heparin; hemostasis; nadroparin; anti-Xa; endogenous thrombin potential
MeSH Terms: conditions — Acute Kidney Injury; Multiple Organ Failure | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hemofiltration at 4L/h (Active Comparator): Hemofiltration was started at 4L/h and crossed over to 2L/h after 60 minutes of hemofiltration
  Interventions: Procedure: CVVH 4 to 2 L/h
- hemofiltration at 2L/h (Active Comparator): hemofiltration was started at 2L/h and crossed over to 4L/h after 60 min
  Interventions: Procedure: CVVH 2 to 4L/h

INTERVENTIONS:
Procedure: CVVH 4 to 2 L/h — CVVH is initiated at 4L/h and is converted to 2L/h after 60 min
  Other Names: continuous venovenous hemofiltration
  Arms: hemofiltration at 4L/h
Procedure: CVVH 2 to 4L/h — CVVH is initiated at 2L/h and is converted to 4L/h after 60 min
  Other Names: continous venovenous hemofiltration
  Arms: hemofiltration at 2L/h

SUMMARY:
The low molecular weight heparin nadroparin is used for anticoagulation of the extracorporeal hemofiltration circuit. Continuous hemofiltration is a renal replacement modality for intensive care patients with acute renal failure. Up to now it is not known whether nadroparin is removed by hemofiltration or not. Accumulation would increase the risk of bleeding.

Aim of the present study is to determine

1. whether nadroparin accumulates in plasma
2. whether nadroparin is removed by filtration and whether removal depends on hemofiltration dose
3. the effects of nadroparin during critical illness on coagulation and anticoagulation

DETAILED DESCRIPTION:
The low molecular weight heparin (LMWH) nadroparin is used for anticoagulation of the extracorporeal hemofiltration circuit. LMWH accumulate in patients with chronic renal failure. Continuous venovenous hemofiltration (CVVH) is a renal replacement modality for intensive care patients with acute renal failure. Up to now it is not known whether nadroparin is removed by hemofiltration or not. If not, accumulation is expected and the risk of bleeding for the patient increases. Because critically ill patients are at increased risk of bleeding, this question is crucial.

If nadroparin would be removed by filtration, removal is expected to depend on hemofiltration dose (to be greater with a higher dose)

We therefore designed a randomized controlled cross-over trial in the setting of critical illness and acute renal failure comparing the anticoagulant effect of nadroparin (anti-Xa) between two doses of CVVH in the patients blood, in the extracorporeal circuit and in the ultrafiltrate.

Because hemostasis in critically ill patients is not only influenced by anticoagulation but also by the critical illness and the extracorporeal circuit, we also measure other hemostatic markers, especially the endogenous thrombin potential (ETP), which seems the most global marker of hemostasis, incorporating procoagulant and anticoagulant effects.

ELIGIBILITY:
Inclusion Criteria:

* acute renal failure requiring renal replacement therapy

Exclusion Criteria:

* (recent) bleeding or a suspicion of bleeding necessitating transfusion,
* need of therapeutic anticoagulation or
* (suspected) heparin-induced thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Accumulation of anti-Xa activity in plasma and removal of anti-Xa activity by filtration. | 24 hours

SECONDARY OUTCOMES:
Endogenous thrombin potential, D-dimers, Prothrombin fragments 1-2, thrombin-antithrombin complexes | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Heleen Oudemans-van Straaten, MD.PhD, Principal Investigator — Onze Lieve Vrouwe Gasthuis
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, Netherlands

REFERENCES:
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078
- [Derived] Oudemans-van Straaten HM, van Schilfgaarde M, Molenaar PJ, Wester JP, Leyte A. Hemostasis during low molecular weight heparin anticoagulation for continuous venovenous hemofiltration: a randomized cross-over trial comparing two hemofiltration rates. Crit Care. 2009;13(6):R193. doi: 10.1186/cc8191. Epub 2009 Dec 3. PMID 19958532